CLINICAL TRIAL: NCT05654207
Title: Answering the Alarm: A System of Care for Black Youth at Risk for Suicide
Brief Title: WeCare: A System of Care for Black Youth
Acronym: WeCare
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH129786-01 (NIH)
Record Dates: First submitted 2022-11-30; First posted 2022-12-16 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-04

CONDITIONS: Suicidal Ideation
Keywords: suicide; ideation; Black youth; depression
MeSH Terms: conditions — Suicidal Ideation; Suicide; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WeCare (Experimental): WeCare system of care - universal screening, ED-based intervention, text message follow-up.
  Interventions: Behavioral: WeCare
- Usual Services (No Intervention): Usual care for youth presenting to the ED will be the control condition.

INTERVENTIONS:
Behavioral: WeCare — WeCare combines two evidence-based strategies -- universal screening using the Computerized Adaptive Screen for Suicidal Youth and an adapted version of the SAFETY-ACUTE, which incorporates PI Lindsey's extensive work with Black youth, their families, and community stakeholders to develop culturally tailored strategies for addressing treatment barriers.
  Arms: WeCare

SUMMARY:
The overall goal of this study is to respond to the urgent need for an effective suicide prevention strategy for Black youth by examining the effectiveness of a systems-level strategy to recognize and respond to suicide risk among Black adolescents who present to emergency departments (EDs). The proposed strategy, WeCare, combines combines three components: (1) universal screening using the Computerized Adaptive Screen for Suicidal Youth (CASSY), (2) a brief intervention designed for Black youth with elevated suicide risk in for ED settings, Connections for Safety (CFS), that combines safety planning and strategies to support linkage to outpatient mental health services, and (3) supportive text messages to youth and parent/caregivers for six weeks following the youth's ED visit. Study objectives are (1) to integrate input from multiple stakeholders to inform and facilitate WeCare implementation, and (2) to use a hybrid one effectiveness-implementation design to evaluate its effectiveness.

DETAILED DESCRIPTION:
From 1991 through 2017, suicide attempts increased by 73% among Black high school-aged youth, and suicide attempts requiring hospitalization increased by 122% for Black high school-aged boys. These alarming findings, in part, led to the creation of the Emergency Taskforce on Black Youth Suicide and Mental Health and their subsequent report, Ring the Alarm: The Crisis of Black Youth Suicide in America, and passage of the Pursuing Equity in Mental Act. These all highlight the urgent need to improve suicide risk detection, treatment, and prevention among Black youth.

We propose to respond to these challenges and the urgent need for an effective suicide prevention strategy for Black youth by examining the effectiveness of an "easily implementable," "systems-level" strategy to recognize and respond to suicide risk among Black youth who present to EDs. WeCare combines (1) CASSY, a universal screening; (2) CFS, an intervention with elements from SAFETY-Acute (SAFETY-A), an evidence-based, family-centered intervention to safety planning for children and adolescents; (3) Safety Planning Intervention (SPI), a brief ED-based intervention of a written list prioritizing coping strategies and sources of support to alleviate a suicidal crisis; (3) Making Connections Intervention (MCI), a mental health engagement intervention for Black adolescents and their parents; and (4) a follow-up text messaging support system for youth and parents will be introduced for enhanced feasibility.

This study is a randomized clinical effectiveness trial with 2,200 Black youth at risk for suicide to examine the effectiveness of WeCare. Youth, ages 12 to 19 years, enrolled from two hospital EDs in New York City, will be assessed on enrollment for risks associated with suicide. Moderate/high-risk youth will be randomly assigned to WeCare vs. usual services. Survey assessments will be conducted at 3- and 6-month follow-up, with medical record review through 12 months to examine the effectiveness of WeCare and mediators of WeCare effects. The objective is to increase risk identification, treatment referral and engagement, and, in turn, reduce suicidal ideation and behavior among Black youth.

ELIGIBILITY:
Inclusion criteria adolescent and parent/guardians:

* Adolescents aged 12-17 years and their parents or guardians, and adolescents 18-19 years who have the option for their parent or guardian to participate
* Having a parent/caregiver present in the ED to consent (12-17 year olds, only)
* Having a cellular phone with text messaging capacity
* Adolescent able to speak English, and understand study questions
* Parents able to consent in English, Spanish, French or Creole
* Meet screening criteria

Exclusion criteria adolescent and parent/guardians:

* Adolescent is medically unstable
* Adolescent present with severe cognitive impairment
* Parents are not present in the ED and available to give consent in either English, Spanish, French or Creole (12-17 year olds, only)
* Adolescent does not have access to cellular phone
* Adolescents active in mental health treatment (e.g., seen a therapist, social worker, or mental health provider in the last week)

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2200 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Mental Health Outpatient Visits (Electronic Medical Record) | Baseline, Months 3 and 6
  This measure assesses mental health service utilization from 50 patient care locations in New York City via electronic medical records.
Columbia-Suicide Severity Rating Scale | Baseline, Months 3 and 6
  This measure is a semi structured interview to assess suicidal ideation and attempt This measure is a semi structured interview to assess suicidal ideation and attempt behavior (actual, interrupted, aborted suicide attempts; preparatory behavior).

SECONDARY OUTCOMES:
Attitudes Toward Psychological Help Scale | Baseline, Months 3 and 6
  This measure assesses psychological factors, including stigma, perceived relevance of treatment, etc. that impact one's perceptions and attitudes about using formal mental health treatment services.
Barriers | Baseline, Months 3 and 6
  This 5-item measure captures barriers to MH treatment participation identified in PI Lindsey's prior work with Black youth and families. A higher score indicates a perception of more barriers to treatment (Minimum score: 5; Maximum score: 15).
Caregiver Knowledge of Mental Health Services (Therapy Survey) | Baseline, Months 3 and 6
  This measures expectations about treatment at a children's psychiatric clinic (caregiver).
ED STARS Mental Health Service Use | Baseline, Months 3 and 6
  This measure assesses mental health service utilization, efforts to link to services, linkage, and engagement with outpatient MH services (caregiver).
Hopelessness | Baseline, Months 3 and 6
  This measure targets recent feelings of hopelessness and hope.
Parent-Family Connectedness Scale | Baseline, Months 3 and 6
  This measure assesses familial connectedness.
How I Feel about Friends | Baseline, Months 3 and 6
  This 2-ite, measure assesses peer connectedness. Higher scores indicate greater peer connectedness (Minimum score: 2; Maximum score: 10).
Peer Victimization and Perpetration | Baseline, Months 3 and 6
  This measure assesses bullying.
Urgency Premeditated Perseverance Sensation Seeking Subscale | Baseline, Months 3 and 6
  This measure assesses impulsivity.
Mental Health Service Use | Baseline, Months 3 and 6
  This measure assesses lifetime mental health service use (caregiver).
Stages of Change | Baseline, Months 3 and 6
  This 8-item measure assesses adolescents' willingness to change (Minimum score: 8; Maximum score: 32).
Barriers to Treatment Participation Scale | Baseline, Months 3 and 6
  This measure assesses barriers to treatment (caregiver).

OTHER OUTCOMES:
Self-Efficacy | Baseline, Months 3 and 6
  This measure assesses adolescents' confidence in use of different coping behaviors (commonly incorporated in safety plans) when experiencing suicidal thoughts.
YRBS-Alcohol | Baseline, Months 3 and 6
  This measure assesses alcohol use.
Drug Use Scale | Baseline, Months 3 and 6
  This measure assesses adolescents' behaviors related to drug use.
YRBS-Physical Fights | Baseline, Months 3 and 6
  This single item measures frequency of physical fighting with a higher score indicating more incifidenst of fighting.
Lethal Means Restriction | Baseline, Months 3 and 6
  This measure assesses adolescents' access to lethal means (caregiver).
Perceived Effectiveness of Treatment | Baseline, Month 3
  This measure assesses perceived treatment effectiveness.
Purpose in Life | Baseline, Months 3 and 6
  This measure assesses adolescents' sense of purpose
Thoughts about Mortality | Baseline, Month 6
  This 5-item measure assesses beliefs and attitudes towards death.
Suicidal Thoughts | Baseline, Months 3 and 6
  This instruments measures the frequency of suicidal thoughts (only if participant responds YES to CSSRS 1 or 2).
Exposure to Suicide | Baseline, Months 3 and 6
  This measure assesses if adolescents had exposure to someone who attempted or died by suicide.
Acquired Capability for Suicide | Baseline, Months 3 and 6
  This 4-item measure assesses fearlessness of death.
Demographics | Baseline, Months 3 and 6
  This survey queries background characteristics (youth and caregiver versions).
Gender Identity and Sexual Orientation | Baseline, Months 3 and 6
  This survey queries adolescents' gender identity and sexual orientation.
Purpose in Life (Expanded) | Months 3 and 6
  Expanded 6-item version of baseline purpose of life measure.
Regard of Identity | Baseline, Months 3 and 6
  This 2-item measure assesses regard for racial identity.
Social Competencies | Baseline, Months 3 and 6
  This 3-item measure assesses social skills.
Religious Identity | Baseline, Months 3 and 6
  This survey queries religious identity (caregiver).
Medical Mistrust | Baseline, Months 3 and 6
  This 5-item measure assesses medical mistrust (caregiver). Higher score sindicate more medical mistrust (Minimum score: 6; Maximum score: 30).
PedsQL | Baseline, Months 3 and 6
  This measure assesses caregiver-reported issues youth face.
ED-s Risk Survey (from ED-STARS) | Baseline, Months 3 and 6
  This survey measure assesses the duration of suicidal thoughts, family and social connectedness, peer victimization and bullying, impulsive-aggression, physical fighting, and overall adaptive functioning.
Work and Social Adjustment Scale - Youth (Parent version) | Months 3 and 6
  This measure assesses the impact of youth's problem to do certain day-to-day tasks (caregiver).
iBelong | Baseline, Month 6
  This 6-item measure assesses adolescents' sense of belongingness. Higher scores indicate greater belongingness (Minimum 6; maximum 30).
Joy | Months 3 and 6
  This 2-item measure assesses adolescents' sense of joy in their life.
Data Archive Collection Items | Baseline, Months 3 and 6
  These items are shared data with the wider scientific community to assess mental and physical health concerns and wellbeing.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Lindsey, PhD, Principal Investigator — New York University
Locations (1):
- Kings County Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Submit data in compliance with NIMH Data Archive data submission agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: By the end of data collection, March 2027.
Access Criteria: In accordance with the NIMH Data Archive requirements.